CLINICAL TRIAL: NCT03252977
Title: The Effectiveness of Tailored Patient Controlled Analgesia Based on Preoperative Pain Sensitivity in Gynecological Patients
Brief Title: Tailored PCA Based on Preoperative Pain Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Associate professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-1707-078-869
Record Dates: First submitted 2017-08-14; First posted 2017-08-17 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Analgesia, Patient-Controlled
Keywords: fentanyl; Pain Threshold; predicted
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tailored group (Experimental): Tailored regimen of IV PCA according to pain sensitivity The regimen of IV PCA will be determined according to preoperative pain sensitivity of patients. Pressure pain threshold will be measured preoperatively in these patients using pressure algometer. Patients with low pain threshold will use high dose IV PCA containing fentanyl 1500mcg, while patients with high pain threshold will use low dose IV PCA containing fentanyl 1000mcg.
  Interventions: Other: Tailored regimen of IV PCA according to pain sensitivity
- control group (Sham Comparator): Regimen of IV PCA without considering pain sensitivity The regimen of IV PCA will be determined according to experimental group patient assignments. Pressure pain threshold will not be measured in these patients. Patients will use IV PCA with fentanyl 1000mcg or fentanyl 1500mcg. The determination will be paired to assignment of experimental group.
  Interventions: Other: Regimen of IV PCA without considering pain sensitivity

INTERVENTIONS:
Other: Tailored regimen of IV PCA according to pain sensitivity — In tailored group, fentanyl dosage in IV PCA will be determined according to preoperative pain sensitivity. In control, group, fentanyl dosage in IV PCA will be determined without consideration of patient's pain sensitivity.
  Arms: Tailored group
Other: Regimen of IV PCA without considering pain sensitivity — In control group, regimen of IV PCA will be determined without consideration about patient's pain sensitivity.
  Arms: control group

SUMMARY:
Opioids via intravenous patient-controlled analgesia (IV PCA) are widely used for postoperative pain control. However, effective pain control with minimized side effects of analgesic agents is still challenging. Several studies reported that preoperative pain sensitivity measured by quantitative sensory test could predict postoperative pain. Therefore, the investigators planned this trial to evaluate the effectiveness of tailored patient-controlled analgesia based on preoperative pain sensitivity measured by pressure pain threshold in patients undergoing gynecological surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled to undergo elective gynecological surgery under general anesthesia
* patients scheduled to use IV PCA for postoperative analgesia
* patients with American Society of Anesthesiologists (ASA) physical status classification I, II, III

Exclusion Criteria:

* contraindication to fentanyl use
* inability to communication
* age less than 18 years, or more than 80 years
* body weight less than 40kg, or more than 90kg
* morbid cardiovascular disease
* pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2017-08-21 (Actual); Primary Completion 2017-11-21 (Actual); Study Completion 2017-11-24 (Actual)

PRIMARY OUTCOMES:
postoperative nausea | during the postoperative 3 days
  Incidence of postoperative nausea

SECONDARY OUTCOMES:
postoperative pain scores | during the postoperative 3 days
  numeric rating scale
incidence of postoperative vomiting | during the postoperative 3 days
  incidence of postoperative vomiting
Severity of postoperative nausea | during the postoperative 3 days
  numeric rating scale
Incidence of other postoperative adverse effects | during the postoperative 3 days
  itching sense, urinary retention, drowsiness, dry mouth, sweating, respiratory depression
cumulative dose of drug that infused via IV PCA | during the postoperative 3 days
  cumulative dose of drug that infused via IV PCA
Incidence of IV PCA clamping | during the postoperative 3 days
  Incidence of IV PCA clamping
rescue analgesics | during the postoperative 3 days
  amount of administered rescue analgesics
antiemetic agents | during the postoperative 3 days
  amount of administered antiemetic agents
satisfaction score | during the postoperative 3 days
  Patient's satisfaction with postoperative analgesia (0:totally unsatisfied and 100: totally satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tae Kim, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahmad S, De Oliveira GS Jr, Bialek JM, McCarthy RJ. Thermal quantitative sensory testing to predict postoperative pain outcomes following gynecologic surgery. Pain Med. 2014 May;15(5):857-64. doi: 10.1111/pme.12374. Epub 2014 Feb 12. PMID 24517836
- [Background] Hsu YW, Somma J, Hung YC, Tsai PS, Yang CH, Chen CC. Predicting postoperative pain by preoperative pressure pain assessment. Anesthesiology. 2005 Sep;103(3):613-8. doi: 10.1097/00000542-200509000-00026. PMID 16129988